CLINICAL TRIAL: NCT03502031
Title: Safety and Efficacy of Maximally Tolerated RAAS Blockade and Spironolactone Therapy on Urinary Proteinuria and Progression of Type II Diabetic Nephropathy in African Americans and Other Patient Cohorts.
Brief Title: Safety and Efficacy of Two Year of RAAS Alone or in Combination With Spironolactone Therapy
Acronym: MRA-ACE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: James A. Tumlin, MD (Other)
Collaborators: Nelson Kopyt, MD (Unknown)
Responsible Party: Sponsor-Investigator, James A. Tumlin, MD, Sponsor-Investigator, NephroNet, Inc.
Organization: NephroNet, Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN-01
Record Dates: First submitted 2017-11-13; First posted 2018-04-18 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Renal Insufficiency, Chronic; Diabetic Nephropathy Type 2
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Single Person; Enalapril; Perindopril; Spironolactone; Lisinopril; Losartan; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- RAAS alone (Active Comparator): RAAS (Lisinopril, Enalapril, Perindopril, Losartan, and Valsartan taken each day at maximum tolerated dose that will different for each subject)
  Interventions: Drug: Renin-Angiotensin (RAAS) alone
- RAAS in Combination with Spironolactone (Active Comparator): RAAS (Lisinopril, Enalapril, Perindopril, Losartan, and Valsartan taken each day at maximum tolerated dose that will different for each subject); Spironolactone taken each day at 25mg
  Interventions: Drug: Renin-Angiotensin (RAAS) blockers in combination with Spironolactone

INTERVENTIONS:
Drug: Renin-Angiotensin (RAAS) alone — maximal RAAS blockade alone for 24months.
  Other Names: Lispril, Enalapril, Perindopril, Losarta, Valsar etc.,
  Arms: RAAS alone
Drug: Renin-Angiotensin (RAAS) blockers in combination with Spironolactone — maximal RAAS blockade alone or in combination with Spironolactone (25 mg) for 24 months.
  Other Names: Lisinopril, Enalapril, Perindopril, Losartan, Valsartan, or Spironolactone
  Arms: RAAS in Combination with Spironolactone

SUMMARY:
NephroNet proposes to examine whether combining Spironolactone with maximal RAAS blockade will further reduce urinary protein at one year and whether prolonged therapy (24 months) is able to slow the decline in GFR. Because of combination MRA and RAAS therapy significantly increases the risk for clinically significant hyperkalemia, we also plan to determine whether the addition of Patiromer to these patients facilitates the use of combination therapy and allows a larger proportion of diabetic patients the potential benefit of combination therapy on renal function.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Male or Female
* Patients with Type II diabetes mellitus must be receiving oral agents or insulin injections at the time of randomization
* All eligible patients will be on a stable, maximum to dose of an ACE or ARB for 2 weeks prior to randomization.
* Note: The determination of m tolerated ACE-ARB therapy will be left to the discretion of the site princ
* All eligible patientswill have hypertension targetblood pressur of < 140/90mm Hg.
* Antihypertensiv therapy may be adjusted to achieve the target blood pressure prior to the time of randomization.
* ACE or ARB therapy will be the primary antihypertensive therapy used for blood pressure control and will be titrthe highest tolerated dose to achieve a target blood pressure of <Patients requiring additional medications to achieve the target blood pressure will use antihypertensive agents that have neutral effects on urinary proteinuria (e.g. Hydralazine or lo Dihydropyridine calcium channel blockers etc.). CcThe final choice of additional medications will be left to the discretion of the site principal investigator (PI)
* Patients with anurine protein to creatinine (UP/Cr) ratio that is mg/gm from the average of two historical value within one year prior to randomization will be considered eligible for study entry.
* Patients with a baseline K+ of >5. X5 meq/l on maximum tolerated ACE-ARB therapy during the screening period can be treated with 8.4 grams of Patiromer for 7 days. If at the end of 7days the serum K+ is < 5.0 meq/liter the patient will be considered eligible to participate in the study. If at the end of 7 days the serum K+ >5.0 meq/l the dose of Patiromer can be increased to 16.8 grams. If at the end of 7 days the serum K+ is < 5.0 meq/L, the patient will be considered eligible for study entry. If after 7 days at the higher dose of Patiromer the serum K+ >5.0, the patient will be ineligible for study participation.
* Patients with an estimated GFR by CK-Epi .73 m2
* Female patients will be required to undergo routine birth control measures

Exclusion criteria:

* Estimated GFR by MDRD20 mls/min/1.73 M2 using the CKD-Epi equation
* Patients with serum K+ > 5.00 while taking 16.8/day of Patiromer
* Patients with history of Type mellitus
* Patients with HgbA
* Pregnant or breast-feeding female patients
* Female patients unwilling to receive estrogen or progesterone based birth control or are unwilling or unable to usconventional barrier birth control methods.
* Patients with known allergy or intolerance tor Spironolactone therapy
* Patients taking oral or IV digoxin
* Patients receiving chronic steroids > 1oral Prednisone
* Patient that do nohave minimum o eGFR determinations within 2 years prior to study randomization
* Concurrent use of Amiloride, , Aliskerin, or other Aldosterone antagonists Patien receiving any of the above medications will be considered eligible for study participation after a wash-out

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Combination Therapy - RAAS inhibition and Spironolactone to lower UP/Cr | 24 months
  To determine whether combination therapy with maximall RAAS inhibition and Spironolactone is superior to RAAS inhibition alone in lowering the UP/Cr ratio at 12 months

SECONDARY OUTCOMES:
Combination Therapy - RAAS inhibition and Spironolactone | 24 months
  To determine whether combination therapy with maximally tolerated RAAS inhibition and Spironolactone is superior to RAAS inhibition alone in slowing the progression of renal disease as evidenced by changes in GFR
Combination Therapy - RAAS inhibition and Spironolactone that develop hyperkalemia | 12 months, 24 months
  To determine the patients in the maximal RAAS blockade group and those receiving combination RAAS + Spironolactone therapy developing clinically significant hyperkalemia as defined as a serum K+ level greater than 5.5 meq/L. We will determine the percentage of patients that require "Patiromer-Rescue" for K+ > 5.5 meq/L and the percentage of patients maintained with serum K+ less than 5.5 meq/L

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Georgia Nephrology Research Institute, Lawrenceville, Georgia
  - Nelson Kopyt, MD, Bethlehem, Pennsylvania

IPD SHARING:
Plan to Share IPD: No